CLINICAL TRIAL: NCT03215485
Title: The WAVE~Ripples for Change: Obesity Prevention in Active Youth in Afterschool Programs Using Virtual- and Real-World Experiential Learning
Brief Title: WAVE~Ripples for Change: Obesity Prevention in Active Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6317
Record Dates: First submitted 2016-05-19; First posted 2017-07-12 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Childhood Obesity Prevention
Keywords: adolescent; sports; nutrition; physical activity; body mass index; virtual world
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: There is one intervention group and one comparison group.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): All intervention youth participants will receive three components:
  1. Nutrition lessons
  2. Virtual World learning environment
  3. Newsletters
  Interventions: Behavioral: Nutrition lessons; Behavioral: Virtual world learning environment; Other: Newsletter
- Comparison (Active Comparator): All comparison youth participants will only receive one component:
  1) Newsletters
  Interventions: Other: Newsletter

INTERVENTIONS:
Behavioral: Nutrition lessons — Face-to-face interactive group lessons delivered in the classroom.
  Arms: Intervention Group
Behavioral: Virtual world learning environment — Every participant has their own unique avatar in the virtual world learning environment named Rippleville. They can choose to complete quests, watch archived nutrition video lessons, explore, and socialize with other avatars. They receive rewards (Rippleville dollar and badges) for their efforts.
  Other Names: Rippleville
  Arms: Intervention Group
Other: Newsletter — All participants in the intervention and comparison groups receive up to 10 professional newsletters on topics related to sports nutrition and performance, healthy eating and active living tips.

SUMMARY:
Intervention targets youth ages 14 - 19 participating in soccer teams. The intervention group will be given face to face nutrition lessons and have access to an online immersive learning environment. The comparison group will not. The project will test if the immersive learning environment is effective in preventing unhealthy weight gain.

DETAILED DESCRIPTION:
Active youth are just as likely to develop poor dietary habits that can contribute to obesity later in life, after high school sports has ended. However, youth in sports may provide a key "window of opportunity" to teach them about eating health foods if that information is tied to sport performance. This project will test to see if that is true.

The virtual world is an idea medium for learning for this project. The project will test whether it indeed can result in behavior change more effectively than just more traditional face to face learning.

ELIGIBILITY:
Inclusion Criteria:

* youth ages 14 - 19 at baseline
* enrolled in a high school soccer program
* living with a parent/caregiver in Oregon
* without medical condition that hinders them from consuming normal healthy diets
* has assess to the internet during the 2-year study
* proficient in English

Exclusion Criteria:

* non-English speakers (youth)
* prisoners

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 498 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Nutrition: Meet specific good groups dietary recommendation/guideline for fruit, vegetables, fat, and sugar intakes. | Change from baseline at 12 and 24 months later
  Intakes of fat, sugar, fruits and vegetables are measured by self-reported screener using the Block Food Frequency Questionnaires (FFQ). Change in intake frequencies are compared baseline, 12 and 24 months later.
Physical activity: Meet moderate to vigorous physical activity (MVPA) recommendation. | Change from baseline at 12 and 24 months later
  MVPA is measured by total steps and minutes per day with the use of a wearable lifestyle tracker such as the Fitbit. Average steps during soccer season and outside soccer season are compared.
Sleep about 8 hours/day. | Change from baseline at 12 and 24 months later
  Together with MVPA, sleep is measured by average number of sleep hours per day as self-reported by participants via written and/or electronic surveys .

SECONDARY OUTCOMES:
Growth-adjusted Body Mass Index (kg/m2) | Change from baseline at 12 and 24 months later
  Height and body weight are measured using a stadiometer (SECA 217, SECA Corp., Singapore) and a Tanita scale (TM-300A, Tanita Corp., Itabashi-Ku, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Overall Officials: Siew Sun Wong, PhD, Principal Investigator — OSU; Melinda M Manore, PhD, RD, Principal Investigator — OSU

IPD SHARING:
Plan to Share IPD: Yes
We will provide IPD (with participant's full name deidentified with a unique ID) upon request after the completion of the study for research and education purpose (not for-profit/commercial use). Types of data available include demography, anthropometry, nutrition, physical activity, sleep, psychosocial, and knowledge in sports nutrition.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will become available in 2019 for up to two years.
Access Criteria: All requests will be sent to the Lead PD (Wong) and approval will be made jointly by both PD Wong & Manore.